CLINICAL TRIAL: NCT06050876
Title: Gallbladder Volvulus Diagnosed Intraoperatively: Case Report
Status: Completed | Type: Observational
Sponsor: University of Balamand (Other)
Responsible Party: Principal Investigator, Omar Tabbikha, General Surgery Resident, University of Balamand
Other Study IDs: UBalamandMLH
Record Dates: First submitted 2023-09-16; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Gallbladder Volvulus
Keywords: Gallbladder volvulus; Acalculous cholecystitis
MeSH Terms: conditions — Acalculous Cholecystitis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Gallbladder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy for gallbladder volvulus — Laparoscopic cholecystectomy for volvulus of gallbladder

SUMMARY:
85-year-old female patient presented with right upper quadrant pain of one day duration, diagnosed with acalculous cholecystitis, and intraoperatively diagnosed with gallbladder volvulus.

DETAILED DESCRIPTION:
85-year-old female patient presented with right upper quadrant pain of one day duration that is associated with nausea and vomiting, but no fever or jaundice. She was tachycardiac and had severe abdominal right upper quadrant tenderness with positive Murphy's sign. Laboratory results showed only increase in inflammatory markers. Both ultrasound and computed tomography scan of the abdomen were done and acalculous cholecystitis was diagnosed. Open cholecystectomy was done but gallbladder volvulus was noted intraoperatively. Cholecystectomy was done and the patient had smooth postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* any patient presenting with right upper quadrant pain

Exclusion Criteria:

* patients having non gallbladder related pathologies explaining right upper quadrant pain

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting with signs and symptoms of a calculus cholecystitis
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Gallbladder volvulus | 1 month
  Intraoperative presence of gallbladder volvulus

CONTACTS AND LOCATIONS:
Locations (1):
- University of Balamand, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
Publishing a case report